CLINICAL TRIAL: NCT00474786
Title: A Randomized Trial Of Temsirolimus Versus Sorafenib As Second-Line Therapy In Patients With Advanced Renal Cell Carcinoma Who Have Failed First-Line Sunitinib Therapy
Brief Title: Temsirolimus Versus Sorafenib As Second-Line Therapy In Patients With Advanced RCC Who Have Failed First-Line Sunitinib
Acronym: INTORSECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-404; B1771003
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic or Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sorafenib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sorafenib
- 2 (Experimental)
  Interventions: Drug: temsirolimus (Torisel)

INTERVENTIONS:
Drug: Sorafenib — Subjects randomized to arm B will take sorafenib 400 mg (2 x 200 mg tablets) PO, BID (total daily dose of 800 mg).
  Arms: 1
Drug: temsirolimus (Torisel) — Subjects randomized to arm A will receive temsirolimus (Torisel) 25 mg via IV infusion once weekly. This infusion is to be administered over a 30-60 minute period. Subjects are to be pre-treated with 25-50 mg IV diphenhydramine (or comparable IV antihistamine) approximately 30 minutes before temsirolimus infusion.
  Arms: 2

SUMMARY:
This is an international, randomized, open-label, outpatient, multicenter study. Subjects will be assigned in a 1:1 ratio to 1 of 2 treatment arms: temsirolimus 25 mg once weekly by intravenous (IV) infusion or sorafenib 400 mg by mouth (PO) twice daily (BID). These investigational drugs will be administered in 6-week cycles for the duration of the study, up to 24 months. Subjects will be stratified by nephrectomy status, duration of response to sunitinib therapy, Memorial Sloan Kettering Cancer Center (MSKCC) prognostic group, and RCC tumor histology.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of mRCC (regardless of histology or nephrectomy status) with well-documented Radiological PD by RECIST criteria or clinical PD as judged by the investigator while receiving first-line sunitinib therapy. Subjects must have at least 1 cycle of sunitinib therapy (minimum of four weeks continuously).
* At time of randomization, at least 2 weeks since prior treatment with sunitinib, palliative radiation therapy, and/or surgery.
* At time of randomization, there must be at least 1 measurable lesion per RECIST. Lesions that have been previously irradiated or embolized cannot be selected as target lesions.

  * More criteria apply

Exclusion Criteria:

* Metastatic CNS from RCC.
* Subjects who discontinued Sutent therapy due specifically to intolerance.
* Prior systemic therapy for mRCC other than sunitinib.
* Active ketonuria, secondary to poorly controlled diabetes mellitus

  * More criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (112):
- United States (22):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Meriden, Connecticut
  - Pfizer Investigational Site, Municie, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
- Argentina (5):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Rosario, Santa Fe Province
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Nueva Cordoba
  - Pfizer Investigational Site, San Miguel de Tucumán
- Australia (7):
  - Pfizer Investigational Site, Kogarah, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, South Brisbane, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Elizabeth Vale, South Australia
  - Pfizer Investigational Site, Woodville South, South Australia
- Austria (2):
  - Pfizer Investigational Site, Vienna, Austria
  - Pfizer Investigational Site, Salzburg
- Canada (11):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Cornwall, Ontario
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Providencia, Santiago Metropolitan, Chile
- Pfizer Investigational Site, Hong Kong, China
- Denmark (2):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Herlev
- Finland (2):
  - Pfizer Investigational Site, Tampere
  - Pfizer Investigational Site, Turku
- France (16):
  - Pfizer Investigational Site, Montpellier, Cedex 5
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Saint Herlain/Nantes Cedex
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Villejuif
- Germany (8):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Neuss
  - Pfizer Investigational Site, Ulm
- Pfizer Investigational Site, Budapest, Hungary
- Italy (5):
  - Pfizer Investigational Site, Chieti
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Roma
- Netherlands (3):
  - Pfizer Investigational Site, Dordrecht
  - Pfizer Investigational Site, Leeuwarden
  - Pfizer Investigational Site, Zwolle
- Pfizer Investigational Site, Singapore, Singapore
- Pfizer Investigational Site, Seoul, South Korea
- Spain (7):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
- Switzerland (7):
  - Pfizer Investigational Site, Kleinriehenstrasse 30, Basel
  - Pfizer Investigational Site, Basel, Canton of Basel-City
  - Pfizer Investigational Site, Geneva, Canton of Geneva
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bruderholz
  - Pfizer Investigational Site, Lucerne
  - Pfizer Investigational Site, Rheinstrasse 26
- United Kingdom (7):
  - Pfizer Investigational Site, Edgbaston, Birmingham
  - Pfizer Investigational Site, Cambridge, Cambridgeshire
  - Pfizer Investigational Site, Withington, Manchester
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] de Velasco G, McKay RR, Lin X, Moreira RB, Simantov R, Choueiri TK. Comprehensive Analysis of Survival Outcomes in Non-Clear Cell Renal Cell Carcinoma Patients Treated in Clinical Trials. Clin Genitourin Cancer. 2017 Dec;15(6):652-660.e1. doi: 10.1016/j.clgc.2017.03.004. Epub 2017 Mar 21. PMID 28410911
- [Derived] Grunwald V, Lin X, Kalanovic D, Simantov R. Early Tumour Shrinkage: A Tool for the Detection of Early Clinical Activity in Metastatic Renal Cell Carcinoma. Eur Urol. 2016 Dec;70(6):1006-1015. doi: 10.1016/j.eururo.2016.05.010. Epub 2016 May 26. PMID 27238653
- [Derived] Hutson TE, Escudier B, Esteban E, Bjarnason GA, Lim HY, Pittman KB, Senico P, Niethammer A, Lu DR, Hariharan S, Motzer RJ. Randomized phase III trial of temsirolimus versus sorafenib as second-line therapy after sunitinib in patients with metastatic renal cell carcinoma. J Clin Oncol. 2014 Mar 10;32(8):760-7. doi: 10.1200/JCO.2013.50.3961. Epub 2013 Dec 2. PMID 24297950
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3066K1-404&StudyName=Temsirolimus%20Versus%20Sorafenib%20As%20Second-Line%20Therapy%20In%20Patients%20With%20Advanced%20RCC%20%20Who%20Have%20Failed%20First-Line%20Sunitinib

RESULTS

PARTICIPANT FLOW:
Groups:
- Temsirolimus: Temsirolimus 25 milligrams (mg) once weekly by intravenous (IV) infusion administered in 6 week cycles for up to 24 months, participants were premedicated with 25-50 mg IV diphenydramine 30 minutes before temsirolimus infusion. In event of toxicity, dose could be modified or held according to the protocol or at the discretion of the investigator.
- Sorafenib: Sorafenib 400 mg (two 200 mg tablets) by mouth (PO) twice daily (BID) administered in 6 week cycles for up to 24 months. In event of toxicity, dose could be modified or held according to the protocol or at the discretion of the investigator.
Period: Overall Study
Arm/Group | Temsirolimus | Sorafenib
Started | 259 | 253
Completed | 0 | 0
Not Completed | 259 | 253
Not completed — Not Meeting Study Criteria | 0 | 1
Not completed — Investigator Request | 2 | 1
Not completed — Death | 189 | 170
Not completed — Discontinuation of Study by Sponsor | 42 | 59
Not completed — Lost to Follow-up | 4 | 7
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 15 | 15
Not completed — Other | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temsirolimus | Sorafenib | Total
Number analyzed (Participants) | 259 | 253 | 512
Age Continuous [Mean (Standard Deviation); unit: years] | 59.96 (10.20) | 59.74 (10.33) | 59.85 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 61 | 127
  Male | 193 | 192 | 385

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Interval from date of randomization until documentation of progressive disease (PD) by an independent tumor assessment according to Response Evaluation Criteria in Solid Tumor (RECIST) or death for any reason whichever occurred first.
Time Frame: Baseline up to 24 Months
Population: Intent to Treat Population (ITT): all randomized participants according to their assigned treatment, regardless of whether they were received any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 259 | 253
months | 4.28 [4.01 to 5.43] | 3.91 [2.80 to 4.21]
Statistical Analysis 1: Comparison: Temsirolimus vs Sorafenib; Test type: Superiority or Other; p = 0.1933, Log Rank — Stratified for nephrectomy status, duration of response to sunitinib therapy, tumor histology, and Memorial Sloan Kettering Cancer Center (MSKCC) prognostic group; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.71 to 1.07] — Hazard ratio less than (<) 1 means temsirolimus (TEMSR) is at lower risk

2. Secondary Outcome: Progression Free Survival (PFS) by Investigator Assessment
Description: Interval from date of randomization until documentation of PD by an investigator tumor assessment, symptomatic deterioration, or death for any reason whichever occurred first.
Time Frame: Baseline up to 24 Months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 259 | 253
months | 5.43 [4.24 to 5.86] | 4.14 [3.26 to 5.36]
Statistical Analysis 1: Comparison: Temsirolimus vs Sorafenib; Test type: Superiority or Other; p = 0.1888, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.70 to 1.07] — Hazard ratio less than (<) 1 means temsirolimus (TEMSR) is at lower risk

3. Secondary Outcome: Percentage of Participants With Tumor Response
Description: Percentage of participants with tumor response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST and evaluated by independent central review. CR/PR persisted on repeat imaging study at least 4 weeks after initial documentation of response. PR had at least 30 percent decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Baseline up to 24 Months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 259 | 253
percentage of participants | 7.7 [4.8 to 11.7] | 7.9 [4.9 to 11.9]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was the duration from randomization to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: Baseline to date of death from any cause (up to 24 months)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 259 | 253
months | 12.27 [10.13 to 14.80] | 16.64 [13.55 to 18.72]
Statistical Analysis 1: Comparison: Temsirolimus vs Sorafenib; Test type: Superiority or Other; p = 0.0144, Log Rank — Stratified for nephrectomy status, duration of response to sunitinib therapy, tumor histology, and MSKCC prognostic group; Cox Proportional Hazard = 1.31, 95% CI 2-sided [1.05 to 1.63] — Hazard ratio <1 means temsirolimus (TEMSR) is at lower risk

5. Secondary Outcome: Percentage of Participants With PFS Events at 12, 24 and 36 Weeks by Independent Assessment
Description: PFS: Interval from date of randomization until documentation of PD by an independent tumor assessment according to RECIST or death for any reason whichever occurred first. PFS calculated as (Weeks)=(randomization date minus first dose date plus 1) divided by 7.
Time Frame: Weeks 12, 24, and 36
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 259 | 253
percentage of participants
  Baseline to Week 12 | 31.2 | 36.7
  Week 13 to Week 24 | 20.9 | 20.1
  Week 25 to Week 36 | 12.3 | 11.2

6. Secondary Outcome: Duration of Response (DR)
Description: Duration of response as defined by the time from CR or PR (whichever status recorded first) until the date of death or PD was objectively documented. Median and its 95 percent confidence interval (95% CI) were estimated using Kaplan-Meier method.
Time Frame: Baseline up to 24 Months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 259 | 253
months | 8.26 [6.71 to 10.36] | 6.96 [4.18 to 17.50]

7. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to 24 months
Population: Safety population: all participants who received at least 1 dose of test article.
Measure: Number; unit: participants
Arm/Group | Temsirolimus | Sorafenib
Number analyzed (Participants) | 249 | 252
participants
  Serious AE | 103 | 86
  Any AE | 248 | 251

ADVERSE EVENTS:
Time Frame: 5.3 years approximately
Description: The same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Temsirolimus | Sorafenib
Serious Adverse Events (participants affected / at risk) | 104/249 | 87/252
Other Adverse Events (participants affected / at risk) | 243/249 | 249/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus (N=249) | Sorafenib (N=252)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Ascites (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oesophageal hypomotility (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4
Asthenia (General disorders) | 3 | 1
Chest pain (General disorders) | 1 | 3
Fatigue (General disorders) | 2 | 4
General physical health deterioration (General disorders) | 8 | 9
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 1 | 2
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 4
Sudden death (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 0 | 1
Cholangitis suppurative (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 2 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 7
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 3
Blood potassium increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 3
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Lung operation (Surgical and medical procedures) | 1 | 0
Medical device implantation (Surgical and medical procedures) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temsirolimus (N=249) | Sorafenib (N=252)
Anaemia (Blood and lymphatic system disorders) | 83 | 34
Lymphopenia (Blood and lymphatic system disorders) | 21 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 5
Diarrhoea (Gastrointestinal disorders) | 74 | 156
Nausea (Gastrointestinal disorders) | 81 | 71
Constipation (Gastrointestinal disorders) | 57 | 55
Vomiting (Gastrointestinal disorders) | 53 | 45
Abdominal pain (Gastrointestinal disorders) | 33 | 41
Stomatitis (Gastrointestinal disorders) | 54 | 18
Abdominal pain upper (Gastrointestinal disorders) | 14 | 25
Dyspepsia (Gastrointestinal disorders) | 15 | 18
Oral pain (Gastrointestinal disorders) | 13 | 5
Fatigue (General disorders) | 99 | 84
Asthenia (General disorders) | 63 | 63
Mucosal inflammation (General disorders) | 74 | 35
Pyrexia (General disorders) | 53 | 28
Oedema peripheral (General disorders) | 57 | 14
Chest pain (General disorders) | 23 | 25
Pain (General disorders) | 20 | 16
Oedema (General disorders) | 17 | 5
Chills (General disorders) | 15 | 6
Nasopharyngitis (Infections and infestations) | 24 | 16
Weight decreased (Investigations) | 35 | 51
Blood creatinine increased (Investigations) | 32 | 6
Aspartate aminotransferase increased (Investigations) | 22 | 15
Blood alkaline phosphatase increased (Investigations) | 26 | 11
Alanine aminotransferase increased (Investigations) | 18 | 17
Blood lactate dehydrogenase increased (Investigations) | 16 | 13
Haemoglobin decreased (Investigations) | 19 | 9
Decreased appetite (Metabolism and nutrition disorders) | 76 | 94
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 53 | 18
Hypercholesterolaemia (Metabolism and nutrition disorders) | 51 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 45 | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 28 | 30
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 29
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 38
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 17
Headache (Nervous system disorders) | 32 | 44
Dizziness (Nervous system disorders) | 20 | 20
Dysgeusia (Nervous system disorders) | 22 | 10
Paraesthesia (Nervous system disorders) | 14 | 10
Insomnia (Psychiatric disorders) | 15 | 16
Anxiety (Psychiatric disorders) | 13 | 7
Dysuria (Renal and urinary disorders) | 13 | 7
Pollakiuria (Renal and urinary disorders) | 13 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 85 | 57
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 67 | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 51 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 19 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 5
Rash (Skin and subcutaneous tissue disorders) | 104 | 87
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 | 131
Pruritus (Skin and subcutaneous tissue disorders) | 63 | 64
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 78
Dry skin (Skin and subcutaneous tissue disorders) | 40 | 36
Erythema (Skin and subcutaneous tissue disorders) | 15 | 29
Nail disorder (Skin and subcutaneous tissue disorders) | 19 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 17
Hypertension (Vascular disorders) | 8 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.